CLINICAL TRIAL: NCT05931315
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy of CaroRite™ on Psychological Well-being, Oxidative Stress and Quality of Life in Healthy Individuals
Brief Title: A Study to Assess the Efficacy of CaroRite™ on Psychological Well-being, Oxidative Stress and Quality of Life in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: BE/230401/CAR/LS
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Psychological Well-Being; Oxidative Stress; Quality of Life
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CaroRite™ (Active Comparator): One capsule to be taken immediately post-dinner / with dinner
  Interventions: Dietary Supplement: CaroRite™
- Placebo (Placebo Comparator): One capsule to be taken immediately post-dinner / with dinner
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: CaroRite™ — One capsule to be taken immediately post-dinner / with dinner
  Arms: CaroRite™
Dietary Supplement: Placebo — One capsule to be taken immediately post-dinner / with dinner
  Arms: Placebo

SUMMARY:
The present study is a randomized, placebo-controlled, double-blind clinical study in which 94 individuals will be screened, and considering a screening failure rate of 20%, approximately 76 participants will be randomized in a ratio of 1:1 to receive either CaroRite™ or placebo and will be assigned a unique randomization code. Each group will have at least 30 completed participants after accounting for a dropout/withdrawal rate of 20%. The intervention duration for all the study participants is 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Male and female individuals aged ≥18 and ≤60 years with low to moderate physical activity level as per International Physical Activity Questionnaire - Short Form (IPAQ - SF).
* BMI of ≥ 25 to ≤ 29.9 kg/m2
* Having at least two of the following five metabolic risk factors:

  1. Waist circumference > 101.6 cm (40 inches) for men and > 88.9 cm (35 inches) for women;
  2. Triglycerides > 150 mg/dL;
  3. Blood pressure ≥ 130 mm Hg (Systolic Blood Pressure) and/or ≥ 80 mm Hg (Diastolic Blood Pressure);
  4. Fasting blood glucose ≥ 100 mg/dL;
  5. low HDL cholesterol level (less than <40 mg/ dL in men and <50 mg/dL in women)
* Individuals with PGWBI scores of moderate distress (between 61 and 72).
* Individuals with history of physical and/or mental exhaustion since last 4 weeks.
* Willing to complete all study procedures including study-related questionnaires and comply with study requirements.
* Willing to abstain from other supplements or medication.
* Ready to give voluntary, written, informed consent to participate in the study.
* No self-reported physical/mental disabilities or gastrointestinal conditions.
* History of stable weight over the last 6 months (<10% change).
* Not currently pregnant, planning to become pregnant, or currently breastfeeding.
* Willing to maintain current dietary and exercise habits, aside from any changes to be made per the study exercise protocol.

Exclusion Criteria:

* Smokers.
* Presence of unstable, acutely symptomatic, or life-limiting illness.
* Individuals with uncontrolled hypertension with systolic blood pressure ≥ 140 mm Hg and diastolic blood pressure ≥ 90 mm Hg.
* Individuals with diagnosed Type II Diabetes Mellitus with FBG ≥ 126 mg/ dL.
* Neurological conditions causing functional or cognitive impairments.
* Unwillingness or inability to be randomized to one of the two intervention groups.
* Hypo- or hyper- thyroidism as assessed by TSH (Thyroid Stimulating Hormone) levels < 0.4 μIU/L and > 4.50 μIU/L.
* Heavy alcohol drinkers defined as follows: For men, consuming more than 4 drinks on any day or more than 14 drinks/week. For women, consuming more than 3 drinks on any day or more than 7 drinks/week.
* History or presence of clinically significant renal, hepatic, endocrine, biliary, gastrointestinal, pancreatic or neurologic disorders that, in the judgment of the Investigator, would interfere with the participant's ability to provide informed consent, comply with the study protocol (which might confound the interpretation of the study results), or put the individual at undue risk.
* Use of any psychotropic medication within four weeks of screening and throughout the study.
* Use of antibiotics or signs of active systemic infection at the time of screening. Treatment visits will be rescheduled to allow the individuals to wash off the antibiotic for at least five days prior to any test visit.
* Use of any supplements (may include probiotics, post-biotics, herbal supplements, synbiotics, enzyme supplements, vitamins with probiotics) within two weeks of screening and throughout the study.
* Individuals that are currently being prescribed (by primary care physician or other health professional) medication or using an over-the-counter product that in the opinion of the study physician will have an effect on food digestion or nutrient absorption during the study.
* Exposure to any non-registered drug product within 3 months prior to the screening visit.
* Unable/unwillingness to complete study specific diaries (digital/paper-based).
* Current use of the following medications: monoamine oxidase inhibitors, prescription or herbal weight loss medications/ dietary supplement.
* Females who are pregnant/planning to be pregnant/lactating or taking any oral contraceptives.
* Individuals with any reported allergy or intolerance to any ingredient in the study products.
* Individuals deemed unsuitable for study based upon study physician assessment.
* Individuals who have been a part of another clinical trial in the past year.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
To assess the impact of the Investigational Product (IP) on psychological well-being using the Psychological General Well-Being Index (PGWBI). | Day 90
  The PGWBI comprises of six sub-scales assessing the positive and negative states on a six-point Likert scale (0 = absence of psychological well-being; to 5 = high levels of well-being). Scores between 0 and 60 indicate severe distress, between 61 and 72 reflect moderate distress, and between 73 and 110 indicate a positive psychological well-being.

SECONDARY OUTCOMES:
Oxidative stress as assessed by decrease in serum levels of 8-Isoprostanes. | Day 90
  The normal reference range of 8-isoprostanes is 2-34 pg/ml
Immune Status as assessed by the increase in salivary IgA levels. | Day 90
  The normal reference range of IgA levels are: male 28.0 - 188.2 ng/ml; female 32.4 - 156.8 ng/ml.
Quality of life as assessed by increase in the scores of SF-36 questionnaire. | Day 90
  The SF-36 includes multi-item scales to measure the following 8 dimensions (refer 15.2 for questionnaire):
  PF- Physical functioning (10 items in question 3) RP- Role limitations due to physical health problems (4 items in question 4) BP- Overall body pain (questions 7 and 8) SF- Social functioning (questions 6 and 10) MH - General mental health, covering psychological distress and well-being (5 items: questions 9 b, c, d, f and h) RE- Role limitations due to emotional problems (questions 5 a, b and c) VT- Vitality, energy or fatigue (4 items: questions 9 a, e, g and i) GH- General health perceptions (5 items: questions 1 and 11 a to d)
Sleep quality as assessed by the decrease in the PSQI score | Day 90
  In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). All the seven component scores are to be added together for calculating the Global PSQI Score. Higher scores indicate worse sleep quality

CONTACTS AND LOCATIONS:
Locations (4):
- India (4):
  - Dr. Praphulla Awate's Clinic, Mumbai, Maharashtra
  - The Kewalramani Clinic, Mumbai, Maharashtra
  - Sangvi Hospital, Pune, Maharashtra
  - Saikrupa Hospital, Pune, Maharashtra

IPD SHARING:
Plan to Share IPD: Undecided